CLINICAL TRIAL: NCT02982525
Title: Effect of Mussel Intake on Vitamin D Status Study
Brief Title: Mussel Intake and Vitamin D Status in Humans
Acronym: Mussel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016/RINH/7
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Disease
Keywords: Mussels; Dietary Intervention; Long-term intervention; Vitamin D status; Selenium; Iodine; Vitamin B12; Omega-3 index
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Mussels (Experimental): The control group will continue to consume their normal habitual diet
  Interventions: Dietary Supplement: No Mussels
- One mussel portion (Experimental): One 75g portion of Scottish mussels provided per week for 12 weeks on top of normal habitual shellfish consumption.
  Interventions: Dietary Supplement: One mussel portion
- Two mussel portions (Experimental): Two 75g portions of Scottish mussels provided per week for 12 weeks on top of normal habitual shellfish consumption
  Interventions: Dietary Supplement: Two mussel portions
- Three mussel portions (Experimental): Three 75g portion of Scottish mussels provided per week for 12 weeks on top of normal habitual shellfish consumption
  Interventions: Dietary Supplement: Three mussel portions

INTERVENTIONS:
Dietary Supplement: No Mussels — Habitual diet only
  Arms: No Mussels
Dietary Supplement: One mussel portion — 1 x 75g mussel portions provided per week
  Arms: One mussel portion
Dietary Supplement: Two mussel portions — 2 x 75g mussel portions provided per week
  Arms: Two mussel portions
Dietary Supplement: Three mussel portions — 3 x 75g mussel portions provided per week
  Arms: Three mussel portions

SUMMARY:
A significant proportion of the United Kingdom population have inadequate levels of vitamin D in their blood. Vitamin D is a fat-soluble vitamin that is essential for the growth and maintenance of healthy bones through increasing dietary calcium absorption within the body. A low vitamin D status has also been associated with other diseases such as osteoporosis, cancer (especially colorectal cancer), cardiovascular disease and type 1 diabetes. Our skin is able to synthesise vitamin D upon exposure to sunlight in summer. If exposure to sunlight is limited, then a dietary supply of vitamin D becomes essential.

However, very few foods contain vitamin D. Among the best dietary sources of vitamin D are oily fish (including salmon, mackerel, herring and trout) and fish oils. Recently, the investigators found that certain shellfish, especially mussels, contain significant amounts of a metabolite of vitamin D, 25(OH)D3. Consumption of this metabolite, as a supplement, has already been shown to improve vitamin D status in humans. Whether consumption of mussels improves vitamin D status is unknown.

In this study the investigators will be looking at whether consumption of 1, 2 or 3 portions of mussels per week for 12 weeks increases vitamin D status in healthy people.

DETAILED DESCRIPTION:
Vitamin D, the main forms being vitamin D2 (ergocalciferol) and D3 (cholecalciferol), is a group of fat-soluble secosteroids which are synthesised from ergosterol in fungi and yeast, or from 7-dehydrocholesterol in humans, animals including fish and plants including microalgae, upon exposure to UV radiation. The metabolically inert vitamin D3 is then converted into 25-hydroxy D3 (25(OH)D3) and subsequently into 1α,25-dihydroxy D3 (1,25(OH)2D3).

A significant proportion of the global population have inadequate vitamin D levels - as defined by a plasma 25(OH)D concentration of <25 nM, - a level where the risk of poor musculoskeletal health appears to increase, which is especially apparent in older children, younger adults, older institutionalised individuals and infants from black and ethnic minority groups. Data from the NDNS and other studies suggest that between 29 and 54% of various population groups in the UK have a serum 25(OH)D concentration < 25 nmol/L in the winter. However, summer synthesis of vitamin D, facilitating maintenance of winter serum 25(OH)D concentration ≥ 25 nmol/L is clearly not occurring for many in the UK population (Consultation on draft SACN Vitamin D and Health report). If there is inadequate vitamin D3 synthesis within the skin, generally caused by limited exposure to sunlight, then a dietary supply of vitamin D becomes essential.

Overall however, very few foods contain vitamin D. Among the best dietary sources of vitamin D are oily fish (including salmon, mackerel, herring and trout) and fish oils, providing up to 20g of vitamin D per 100 g. Lower amounts of vitamin D are present in red meat, liver and egg yolks (approximately 1-5g/100 g). Vitamin D in these foods and in fish is primarily in the form of vitamin D3 and its metabolite 25(OH)D3.

Recently, investigators have found that certain shellfish, especially mussels, contain significant amounts of 25(OH)D3, ranging from 0.7 to 9.9 µg/100 g wet weight. Thus far, food composition databases give either very low or no values for levels of vitamin D in shellfish. The amount of vitamin D3 in mussels is either reported to be below the detection limit, or is not analysed, in mussels in the food database analysis. The importance of finding 25(OH)D3 rather than vitamin D3 in mussels is illustrated by the fact that this metabolite is considered 5 times more effective in raising serum 25(OH)D3 levels in humans, and thus vitamin D status, than vitamin D3 itself. An interesting parallel with meat appears. Meat contains little native vitamin D but as better measurement techniques detected more metabolites of vitamin D, which were considered to be more potent, these have been added to food composition tables. Indeed, the apparent increase in vitamin D intakes in the British household food data, in 1995 and 1996, is a direct result of including the potency factor for meat. Taking account of this potency factor, mussels could provide up to 50g of vitamin D per 100g. Whether consumption of mussels improves vitamin D status in humans is however, not known.

According to exploratory meta-regression analyses of RCT data in a number of European (51-60°N) winter-based, dose-related RCTs which used supplemental doses of vitamin D between 0-20 μg/d, have reported vitamin D-serum 25(OH)D concentration slope estimates of 1.55-2.43 nmol/L increment per 1 μg vitamin D (Consultation on draft SACN Vitamin D and Health report). Thus 1, 2 and 3 portions of mussels per week, providing the equivalent of approx. 2.7, 5.4 and 8.0 mg/day (including the potency factor of 5) may increase serum levels of 25(OH)D3 by 4.2-6.6 nmol/L for 1 portion of mussels per week, 8.4-13.1 nmol/L for 2 portions per week or 12.4-19.4 nmol/L for 3 portions of mussels per week

ELIGIBILITY:
Inclusion Criteria:

* BMI ranging from 18-35
* Not having any food allergies
* Not taking any fish oil or certain nutritional / vitamin supplements
* Non-smoker

Exclusion Criteria:

* Regularly take aspirin or aspirin-containing drugs
* Taking drugs or herbal medicines known to alter the haemostatic system in general
* Taking certain dietary supplements / multivitamin tablets
* Anyone suffering from diabetes, hypertension, renal, hepatic or haematological disease
* Heart / circulation problems
* Eating disorders
* Smoking
* Any existing shellfish allergy
* Having difficult venous access or problems giving blood in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Vitamin D status | At baseline and after 12 weeks mussel supplementation
  Serum Vitamin D status will be assessed by measuring plasma 25-hydroxy vitamin D3 by Liquid Chromatography/Mass Spectrometry, the gold standard method

SECONDARY OUTCOMES:
Vitamin B12 status | At baseline and after 12 weeks mussel supplementation
  Vitamin B12 status will be measured in plasma using the microbiological assay using L. Delbrueckii. Lactis
Change in omega-3 index | At baseline and after 12 weeks mussel supplementation
  The Omega-3 index will be measured by Gas Chromatography-Mass Spectrometry. An optimal target level of the Omega-3 index is 8%, and an undesirable level is less than 4%, with 4-8% being an intermediate-risk zone.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje De Roos, PhD, Principal Investigator — University of Aberdeen, The Rowett Institute
Locations (1):
- University of Aberdeen, The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No